CLINICAL TRIAL: NCT07017738
Title: Effect of Neural Mobilization in Upper Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Essam Ahmed Abdelbaky Abdelbaky, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005577
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Upper Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural mobilization + Corrective exercises (Experimental): They will receive neural mobilization in addition to corrective exercises for UCS, 3 times per week for 6 weeks.
  Interventions: Other: Corrective exercises; Other: Neural mobilization
- Corrective exercises (Active Comparator): They will receive corrective exercise for UCS, 3 times per week for 6 weeks.
  Interventions: Other: Corrective exercises

INTERVENTIONS:
Other: Corrective exercises — The corrective exercise program will include various positions: in standing, scapular retraction and arms overhead; in sitting, chin tuck and thoracic extension; in supine, arms in a W shape and horizontal abduction with external rotation; in side-lying, forward flexion starting with arms parallel to the body; and in prone, scapular retraction and depression in a T shape, extension from 90° forward flexion, and horizontal abduction at 90° with external rotation. Exercises will start with three repetitions held for 10 seconds and progress to six repetitions held for 25 seconds, based on overload principles and individual needs. Participants experiencing pain may stop and rest until symptoms subside.
Other: Neural mobilization — Median nerve mobilization will be performed with the patient in a supine position, shoulder abducted to 90°, elbow flexed at 90°, and both wrist and head in a neutral position. The therapist will mobilize the nerve by extending the elbow to 45°, while the patient performs ipsilateral cervical lateral flexion to unload the nervous system.
  Arms: Neural mobilization + Corrective exercises

SUMMARY:
The purpose of this study is to investigate the effect of Neural Mobilization in patients with Upper Cross Syndrome.

DETAILED DESCRIPTION:
Upper cross syndrome (UCS) is the tightness of the levator scapulae, pectoralis major, and upper trapezius whereas inhibition of serratus anterior, deep neck flexors more specifically scalene, middle trapezius, lower trapezius, and rhomboids. This condition is given its name because a cross can be drawn across the upper body. One arm of the cross indicates the tight muscles and the other arm of the cross indicates the inhibited muscles.

People suffering from UCS present with a forward head posture (FHP), hunching of the thoracic spine (rounded upper back), elevated and protracted shoulders, scapular winging, and decreased mobility of the thoracic spine. Sometimes, manual work can cause musculoskeletal disorders, for example, the workers who do their work in awkward positions repeat the same action throughout their workday.

It was found that UCS causes pain among 24.3% of drivers. Also, 35.9% of office workers suffer from the upper cross syndrome and body posture was the leading cause. Housewives were also suffering from upper cross syndrome. The reason behind this is that during household tasks they don't keep a good posture which causes them pain and other difficulties.

Patients complaining of non-traumatic neck pain tend to keep the forward head posture, when compared to people without pain.

Rounded shoulder has been identified as a leading cause of upper quarter pain. Kyphosis, by both clinical and quantitative assessment, causes diminished function especially in tasks that require mobility.

The effect of neural mobilization in various diseases and conditions includes increasing nerve conduction and functional status, decreasing pain and subjective symptoms.

Accordingly, there are no available studies in the literature investigating the effect of neural mobilization on the upper cross syndrome, therefore this is the purpose of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 20 to 50 years.
* Body Mass Index ≤30 kg/m².
* All participants have a forward head, craniovertebral angle < 50°.
* All participants have round back (kyphosis angle ≥ 42°).
* All participants have rounded shoulders of ≥ 52°.
* The subjects were chosen from both genders based on an assessment of upper cross syndrome by photogrammetric analysis.
* All participants have pain intensity level measured by visual analogue scale (4-8).
* All participants tested positive for upper limb tension test of median nerve.

Exclusion Criteria:

* History of trauma or surgery in the cervical region.
* Bone fractures or acute soft tissue injuries.
* Osteoporosis.
* Pregnant women.
* Cancer.
* Neurological conditions affecting cervical and thoracic spine.
* Connective tissue disease: This includes diseases such as osteomyelitis, lupus, and scleroderma.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Forward head angle | 6 weeks
  The forward head angle between the line connecting the tragus and C7 with the perpendicular line will be measured for all participants in both groups pre- and post-treatment, using the photogrammetric method.
Rounded shoulder angle | 6 weeks
  The rounded shoulder angle between the line between the acromion process and C7 with the perpendicular line will be measured for all participants in both groups pre- and post-treatment, using the photogrammetric method.
Kyphosis angle | 6 weeks
  For the kyphosis angle, the bone marker on the spinous process of C7 will be used as the starting point of the arch and the spinous process of T12 will be used as the endpoint of the arch. It will be measured for all participants in both groups pre- and post-treatment, using the photogrammetric method.

SECONDARY OUTCOMES:
Boston Questionnaire (Arabic version) | 6 weeks
  The Boston Questionnaire is a patient-reported outcome measure that has demonstrated reliability, validity, and responsiveness to both surgical and non-surgical treatments. The Arabic version has also been shown to be reliable and valid among Arabic-speaking patients. The questionnaire consists of two separate scales: the Symptom Severity Scale (SSS), which includes 11 questions, and the Functional Status Scale (FSS), which includes 8 items. Respondents rate the difficulty of each item using a five-point scale. Higher scores indicate greater symptom severity or functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Abdelrahman, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt